CLINICAL TRIAL: NCT07151131
Title: Cartoons and Reflexology for Postoperative Nausea, Pain, and Anxiety in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Hava Tetik Özel
Record Dates: First submitted 2025-07-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Children; Pain Management; Nausea, Postoperative
MeSH Terms: conditions — Agnosia; Postoperative Nausea and Vomiting | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Watching Cartoons and Reflexology Massage
  Interventions: Other: Watching Cartoons; Other: Reflexology
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Other: Watching Cartoons — Cartoon Group Intervention Children assigned to the cartoon group will be taken from the clinic to the preoperative room. Approximately 30 minutes before being transferred to the operating room, children will be allowed to watch a cartoon of their choice on a 60-inch screen TV placed approximately 200 cm away. The duration of the cartoon viewing session will be limited to 20 minutes.
  The measurement tools used in the study will be administered at five different time points:
  Immediately before watching the cartoon,
  Immediately after watching the cartoon but before being transferred to the operating room,
  In the postoperative period at the 60th minute,
  At the 120th minute postoperatively,
  And finally, at the discharge phase.
  Arms: intervention group
Other: Reflexology — Massage Group Intervention Children assigned to the massage group will be transferred from the clinic to the preoperative room. Approximately 30 minutes before being taken to the operating room, reflexology massage will be applied by the researcher physician Xxx XXXXX, who holds a valid reflexology certification. The massage will be administered to both the right and left feet, with 10 minutes per foot, for a total duration of 20 minutes.
  The measurement tools used in the study will be applied at five distinct time points:
  Before the massage,
  Immediately after the massage but before operating room transfer,
  In the postoperative period at the 60th minute,
  At the 120th minute postoperatively,
  And finally, during the discharge phase.
  Arms: intervention group

SUMMARY:
Preoperative anxiety arises as a physiological response of the body to stressors and is pathophysiologically associated with stimulation of the autonomic nervous system and increased catecholamine release (Durgut, 2021). As a result, elevated levels of cortisol and epinephrine in the body can cause cytotoxic effects at the cellular level. This physiological mechanism may lead to hypertension, arrhythmia, tachycardia, and tachypnea in children (Dehghan et al., 2019; Durgut, 2021).

Due to these effects, recent evidence-based studies have focused on the use of non-pharmacological approaches with fewer side effects to manage anxiety in children (Kavak et al., 2019). According to the literature, various techniques have been identified as effective interventions for reducing preoperative anxiety in children, including:

Listening to music,

Playing games,

Using dramatic puppets,

Interactive play,

Virtual reality applications,

Watching cartoons,

Playing favorite video games,

Video presentations,

Hospital clowns,

Storybooks,

Visual and auditory stimuli

ELIGIBILITY:
Inclusion Criteria

Participants were included in the study if they met all of the following conditions:

The child was hospitalized in the pediatric surgical clinic for a planned (elective) surgery,

The child was aged between 4 and 6 years,

The child was scheduled to receive general anesthesia,

Neither the child nor the primary caregiver had any visual, hearing, or cognitive impairments,

The child had no anatomical abnormalities or tissue integrity issues in the feet,

Verbal assent was obtained from the child,

Both parents provided written and verbal informed consent for participation,

Both the child and parents were willing and voluntarily agreed to participate in the study.

Exclusion Criteria

Participants were excluded from the study if any of the following conditions occurred:

Postoperative bleeding tendency developed in the child,

The child required postoperative intensive care,

A high-risk complication developed after surgery,

The child failed to initiate spontaneous respiration postoperatively,

Intraoperative death (exitus) occurred,

The child experienced prolonged unconsciousness due to anesthesia,

The child underwent surgical procedures involving the feet.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety Tool: Preoperative Anxiety Scale | Baseline, Postoperative 60th and 120th minutes
Pain Tool: Wong-Baker FACES Pain Rating Scale | Postoperative 60th and 120th minutes
Nausea Tool: standardized observational nausea scale | Postoperative 60th and 120th minutes

IPD SHARING:
Plan to Share IPD: No
Ethically, patient information can be shared upon reasonable request without revealing their identities for security reasons.